CLINICAL TRIAL: NCT05552742
Title: Comparison of The Effects of Virtual Balance Training and Conservative Rehabilitation Therapy on Balance in Stroke Patients.
Brief Title: Comparison of The Effects of Virtual Balance Training and Conservative Rehabilitation Therapy in Stroke Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Abant Izzet Baysal University (Other)
Responsible Party: Principal Investigator, Serdar Kilinc, Assistant Professor, Abant Izzet Baysal University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: AIBU-FTR-SK-04
Record Dates: First submitted 2022-09-21; First posted 2022-09-23 (Actual); Last update posted 2022-09-23 (Actual); Status verified 2022-09

CONDITIONS: Hemiplegia; Stroke
MeSH Terms: conditions — Hemiplegia; Stroke

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conservative Rehabilitation (Active Comparator): Only conservative rehabilitation treatment was applied to the patients in group 1.
  Interventions: Other: Conservative rehabilitation
- Conservative Rehabilitation + Virtual Balance Training (Experimental): Conservative rehabilitation treatment and virtual balance study were applied to the patients in group 2.
  Interventions: Other: Conservative rehabilitation; Device: Virtual Balance Training

INTERVENTIONS:
Other: Conservative rehabilitation — The conservative rehabilitation program includes a patient-specific conservative exercise program comprising exercises that strengthen the paralyzed side, increase joint range of motion and strengthen muscles, stretch spastic muscles, and ensure balance rehabilitation that enhances balance performance and coordination. The patients in both groups received conservative rehabilitation program for 8 weeks, 4 days a week for 1 h.
Device: Virtual Balance Training — Virtual balance training program using the Thera-Trainer Balo device was applied 4 times a week for a total of 8 weeks, and each session lasted for 20 min. The center of mass of each patient was determined using sensors and displayed on the screen. The patients were encouraged to move their mass by swiping in all directions via the apple picking game displayed on the screen
  Arms: Conservative Rehabilitation + Virtual Balance Training

SUMMARY:
The study aimed to assess the effects of a virtual balance training program using the Thera-Trainer Balo (TTB) device along with conservative rehabilitation program on the clinical findings; standing, stepping, walking and balance measures; and activities of daily living in patients with stroke.

DETAILED DESCRIPTION:
Stroke is one of the leading causes of death and disability worldwide. Approximately 71% of stroke cases occur as a result of ischemic infarcts. Most survivors of stroke experience gait and balance disorders that increase the risk of falling.

It has been shown that the functional recovery of patients with stroke is adversely affected and length of hospital stay during the rehabilitation program, particularly in those with severe balance disorders.

Virtual reality technologies are currently employed to accelerate functional recovery in patients.

A total of 30 patients were included in the study. The patients were randomized into two groups with 15 patients in each group by simple randomization.

Group 1 received the conservative rehabilitation program, whereas Group 2 received a balance training program using the Thera-Trainer Balo (TTB) device along with the conservative rehabilitation program.

Patient information regarding the age, gender, hemiplegic side, stroke duration, and type of ischemia were recorded. The stage of motor recovery according to Brunnstrom, spasticity based on the modified Ashworth scale, ambulation ability based on the Functional Ambulation Scale (FAS), quality of life based on the Short Form-36 (SF-36) scale, and balance-coordination status based on the Berg Balance Scale (BBS) were assessed at the beginning of the treatment and at the endpoint of the 8 week treatment. Moreover, evaluations were made with static and dynamic postural stability tests.

The study aimed to assess the effects of a virtual balance training program using the Thera-Trainer Balo (TTB) device along with conservative rehabilitation program on the clinical findings; standing, stepping, walking and balance measures; and activities of daily living in patients with stroke.

ELIGIBILITY:
Inclusion Criteria:

* patients who had a cerebrovascular accident at least 6 months before the study,
* patients had the first unilateral hemiparesis attack, could stand with or without assistance,
* patients had no contraindications for walking.

Exclusion Criteria:

* patients with a history of neurological diseases,
* a mini-mental test score of <24,
* severe spasticity at the lower extremity with grade 4 and unilateral neglect, and musculoskeletal diseases such as amputation and severe arthritis, which limits walking,

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2021-11-01 (Actual); Primary Completion 2022-05-01 (Actual); Study Completion 2022-05-01 (Actual)

PRIMARY OUTCOMES:
Berg Balance Scale | Before Treatment
  The BBS is used to objectively determine a patient's ability to balance safely during a predetermined set of tasks. The scale comprises 14 items. Each item receives a score ranging from 0 to 4, which is a five-point rank scale with 0 indicating the lowest level of functioning and 4 indicating the highest level of functioning
Berg Balance Scale | 8 Week After Treatment
  The BBS is used to objectively determine a patient's ability to balance safely during a predetermined set of tasks. The scale comprises 14 items. Each item receives a score ranging from 0 to 4, which is a five-point rank scale with 0 indicating the lowest level of functioning and 4 indicating the highest level of functioning
Functional Ambulation Scale | Before Treatment
  Functional Ambulation Scale is a 6-point functional walking test that evaluates ambulation ability and determines the amount of human support required by patients while walking, regardless of whether they use a personal assistive device. A score of 0 indicates that the patient has a dysfunctional ambulation A score of 5 denotes independent ambulation on any surface.
Functional Ambulation Scale | 8 Week After Treatment
  Functional Ambulation Scale is a 6-point functional walking test that evaluates ambulation ability and determines the amount of human support required by patients while walking, regardless of whether they use a personal assistive device. A score of 0 indicates that the patient has a dysfunctional ambulation A score of 5 denotes independent ambulation on any surface.
Static and Dynamic Postural Stability Tests | Before Treatment
  In the static postural stability test, two-legged standing, tandem standing, two-legged standing on a foam mat, tandem standing on a foam mat, one-legged standing, turning head and stopping on one leg, and one-legged standing on a foam mat were evaluated. The tasks of walking 25 steps on a foam mat and walking 25 steps on hard smooth ground were evaluated in dynamic postural stability test.
Static and Dynamic Postural Stability Tests | 8 Week After Treatment
  In the static postural stability test, two-legged standing, tandem standing, two-legged standing on a foam mat, tandem standing on a foam mat, one-legged standing, turning head and stopping on one leg, and one-legged standing on a foam mat were evaluated. The tasks of walking 25 steps on a foam mat and walking 25 steps on hard smooth ground were evaluated in dynamic postural stability test.

SECONDARY OUTCOMES:
Brunnstrom Stages | Before Treatment
  Brunnstrom stages is a scale used to assess motor recovery after a stroke, which is expressed using values between 1 and 6. The higher the value on this scale, the higher would be the recovery.
Brunnstrom Stages | 8 Week After Treatment
  Brunnstrom stages is a scale used to assess motor recovery after a stroke, which is expressed using values between 1 and 6. The higher the value on this scale, the higher would be the recovery.
The Modified Ashworth Scale | Before Treatment
  The modified Ashworth Scale is used to evaluate spasticity in patients after stroke, which is expressed using values between 0 and 4. The higher the value on this scale, the higher would be the spasticity.
The Modified Ashworth Scale | 8 Week After Treatment
  The modified Ashworth Scale is used to evaluate spasticity in patients after stroke, which is expressed using values between 0 and 4. The higher the value on this scale, the higher would be the spasticity.
Short Form-36 Quality of Life Scale | Before Treatment
  It consists of 36 questions filled by the individual himself. High scores indicate good quality of life.
Short Form-36 Quality of Life Scale | 8 Week After Treatment
  It consists of 36 questions filled by the individual himself. High scores indicate good quality of life.

CONTACTS AND LOCATIONS:
Locations (1):
- Abant Izzet Baysal University, Bolu, Turkey (Türkiye)